CLINICAL TRIAL: NCT05854979
Title: Ultrasound Assessment of Preoperative Gastric Volume in Fasted, Diabetic Surgical Patients: A Prospective Observational Cohort Study on the Effects of GLP-1 Agonists on Gastric Emptying
Brief Title: Effects of GLP-1 Agonists on Gastric Volume
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Christopher Wolla, Principal Investigator, Assistant Professor, Medical University of South Carolina
Other Study IDs: Pro00128783
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Diabetes; Gastric Content Aspiration; Glucagon-like Peptide 1; GLP-1
MeSH Terms: conditions — Diabetes Mellitus; Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics taking a GLP-1 receptor agonist
  Interventions: Diagnostic Test: Gastric Ultrasound
- Diabetics not taking a GLP-1 receptor agonist (control)
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — A gastric ultrasound will be completed on every patient and administered the same way in each arm. The patient will be placed in supine position. A curvilinear ultrasound probe will be placed on the sagittal plane below the xiphoid process. The probe will then slide along the costal margin to the right until the gastric antrum is identified. At this point, the ultrasound image will be obtained, and appropriate measurements will be taken. The patient will be placed in the right lateral decubitus position and the above procedure will be repeated.

SUMMARY:
This study will enroll patients ages 18 and over who have a diagnosis of diabetes, are undergoing an elective surgery under general anesthesia and 1) are taking a GLP-1 receptor agonist medication, or 2) not taking a GLP-1 receptor agonist medication. The patients will have a gastric ultrasound prior to surgery to measure any retained gastric contents. The primary goal is to assess the effect of subcutaneous injectable GLP-1 agonists on preoperative gastric volume in fasted, diabetic surgical patients.

ELIGIBILITY:
Inclusion Criteria

* Age greater than or equal to 18 years old
* Diagnosed with diabetes (listed on medical record, Hgb A1C greater than or equal to 6.5%, fasting blood glucose greater than or equal to 126mg/dL, and/or on medical treatment for diabetes)
* One of the following groups:
* Taking a GLP-1 Medication
* Not taking a GLP-1 Medication
* ASA Physical Classification Status 1-3
* Scheduled for elective surgery under general anesthesia
* Appropriately fasted per ASA Fasting Guidelines 201712

Exclusion Criteria

* BMI greater than 40
* Previous gastric/esophageal surgery
* Abnormal gastric anatomy
* Pregnancy
* Inability or unwillingness of subject to give informed consent
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of patients with a diagnosis of diabetes who are or are not taking a GLP-1 medication, have appropriately fasted, and scheduled for an elective surgery with general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Gastric Volume in RLD Position | From time of enrollment until the start of surgery, assessed up to 4 weeks
  The gastric volume will be calculated using a validated formula.

SECONDARY OUTCOMES:
Gastric antrum CSA in RLD position | From time of enrollment until the start of surgery, assessed up to 4 weeks
Perlas antral grade | From time of enrollment until the start of surgery, assessed up to 4 weeks
Incidence of aspiration | From the time surgery begins until the end of scheduled surgery, assessed up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wolla, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States